CLINICAL TRIAL: NCT03397472
Title: Magnetic Field Modulation Pillow for Insomnia Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GDREC2017326H(R1)
Record Dates: First submitted 2018-01-04; First posted 2018-01-12 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2018-12

CONDITIONS: Insomnia
Keywords: Insomnia; Treatment; magnetic field modulation
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): use the sleep pillow with the magnetic field modulation treatment
  Interventions: Device: magnetic field modulation device
- placebo group (Placebo Comparator): use the sleep pillow without magnetic field modulation treatment
  Interventions: Device: placebo device

INTERVENTIONS:
Device: magnetic field modulation device — use the device with magnetic field modulation to treat insomnia
  Arms: treatment group
Device: placebo device — use the sleep pillow without magnetic field modulation treatment
  Arms: placebo group

SUMMARY:
This interventional study was designed to explore the clinical effect of magnetic field modulation system on insomnia patients and provide a new solution for insomnia treatment.

DETAILED DESCRIPTION:
Patients with insomnia receiving this sleep pillow with magnetic system or not would be observed in months.The effect of sleep pillow with magnetic system for insomnia would evaluated.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 65 years old. 2.Primary Insomnia

Exclusion Criteria:

1. Secondary Insomnia
2. Pilot, high-altitude operator
3. Pregnant, lactating women
4. Patients with serious disease
5. The researchers believe that the candidates are not eligible

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 5 weeks
  The Sleep Quality of Patients with insomnia as Reflected by PSQI scale.The PSQI scale, consisting of 18 self-rated items, was used to assess the subjects' sleep quality in the last month.The 18 self-rated items can be combined into seven factors: sleep quality, time to fall asleep, sleep duration, sleep efficiency, sleep disorders, hypnotic drugs, and daytime function.Each factor was scored on a scale of 0-3, and the total score of each factor was the total score of PSQI, with the total score ranging from 0-21. The higher the score was, the worse the sleep quality was
Insomnia severity index | 5 weeks
  The severity of insomnia was graded by ISI score，The total score of ISI was 8-14 for mild insomnia, 15-21 for moderate insomnia and 22 for severe insomnia.

SECONDARY OUTCOMES:
Parameters of sleep diary | 5 weeks
  Some parameters of sleep diary
Response rate | 5 weeks
  The total score of Insomnia severity index (ISI) decreased by 50% compared with that before treatment or less than 9 points after treatment will be judged to be responsive. Total number of responsive subject after observation/total number of subject in the group*100%= response rate
Remission rate | 5 weeks
  The total score of Insomnia severity index (ISI) less than 9 points after treatment will be judged to be remissive. Total number of remissive subject after observation/total number of subject in the group*100%= remission rate

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Ou, M.D., Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Genereal Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Previous research plan submitted to the Ethics Committee has stated the participant information not be shared